CLINICAL TRIAL: NCT06139224
Title: Gut Microbiota-Mediated Inflammatory Interactions Between Alcohol Use Disorders and HIV Infection
Brief Title: Gut Microbiota-Mediated Inflammatory Interactions Between AUD and HIV Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Professor, Director of Center for Integrated Microbiome and Chronobiology Research, Rush University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22112903
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder; Human Immunodeficiency Virus
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV-infected ART-suppressed individuals with AUD (Experimental): Only 10 HIV+ ART+,AUD + individuals will be invited to take part in a prebiotic sub study, which they will take a commercially available prebiotic (FOS) for 10 days
  Interventions: Dietary Supplement: 10 day prebiotic consumption
- HIV-infected ART-suppressed individuals with no AUD (Experimental): Only 10 HIV+ ART+,AUD - individuals will be invited to take part in a prebiotic sub study, which they will take a commercially available prebiotic (FOS) for 10 days
  Interventions: Dietary Supplement: 10 day prebiotic consumption

INTERVENTIONS:
Dietary Supplement: 10 day prebiotic consumption — 20 HIV-infected ART-suppressed individuals will be provided a with commercially available prebiotic (FOS) for 10 days. Participants will be instructed to consume the prebiotic daily during the first three days and then twice daily for an additional seven days. Participants will be instructed to consume the powder in the morning on the first three days, then in the morning and afternoon for the following week. Each participant will have a baseline visit and a follow up visit after 10 days of the FOS intervention. Blood and stool will be collected at both visits.

SUMMARY:
Alcohol use disorder (AUD) has been associated with high prevalence of inflammation-associated co-morbidities in people living with HIV even those receiving effective antiretroviral therapy (ART). Our preliminary data support a model in which the combined insult of AUD and HIV on the gut, specifically on the microbiota and intestinal barrier integrity, exacerbates inflammation. Our preliminary data using intestinal organoids also suggest a potential mechanism for AUD-mediated changes in the gut barrier function during HIV; the intestines of HIV+ individuals have low resilience to alcohol induced intestinal barrier disruption caused by high levels of oxidative stress. Finally, our preliminary data also suggest a potential approach to enhance the integrity of the intestinal barrier and reduce gut derived inflammation in people living with HIV with/without AUD- short chain fatty acid prebiotics. These prebiotics prevent alcohol mediated adverse effects on the intestinal barrier and inflammation by preventing oxidative stress. These prebiotics are safe and decrease gut inflammation in humans.

20 HIV+ ART+ (10 AUD- and 10 AUD +), will be recruited for a prebiotic intervention. This is a proof-of-concept observational study to establish a causal link between microbiota-gut and HIV pathology during ART by asking whether modifying microbiota and gut milieu impacts intestinal barrier function, systemic inflammation, and brain pathology in HIV+ people. Participants will have two study visits, where stool collection and blood draw will be collected, as well as questionnaires. These participants are part of the larger observation study (n=160), which will test the hypothesis that intestines from HIV+ individuals have lower resilience to alcohol mediated gut barrier disruption than intestines from HIV-negative controls. We will recruit the following groups of participants: HIV+ ART+ AUD-; HIV+ ART+ AUD+; HIV- AUD- ; HIV- AUD+. Blood, urine, stool, and intestinal biopsies will be collected from participants to compare intestinal barrier integrity, system and gut inflammation, immune activation, oxidative stress, microbiome/metabolome. and HIV reservois. Second, lleal/colonic organoids from HIV- and HIV ART+ individuals will be generated to examine their resilience to alcohol-induced intestinal barrier disruption.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ Group :
* Age 45 to 80 years
* Infection with HIV-1, as documented by a licensed ELISA and confirmed by a Western blot or HIV-1 RNA
* On ART for at least 12 months
* No change in ART for at least three months
* CD4+ T cell count of 350 cells/µl
* Plasma HIV-1 RNA level consistently below the limit of detection of commercial ultrasensitive assays for at least six months before study entry.
* Ability and willingness to provide informed consent
* HIV Negative Group:
* Age 45 to 80 years
* Matched to the HIV+ ART-treated group (age (+/- 5 years), gender, ethnicity, sexual orientation, smoking, and body mass index (+/-3)).
* Ability and willingness to provide informed consent

Exclusion criteria:

* Any condition that, in the opinion of the gastrointestinal (GI) specialist, would either be a contraindication to endoscopy or would increase the risk from sedation, endoscopy, or mucosal biopsies. These conditions may include, but are not limited to:
* Significant complication (such as perforation) from prior endoscopy
* Known bleeding diathesis
* Platelet count < 100,000 per µl
* INR > 1.3
* Current use of antiplatelet agents (aspirin, other NSAIDs, clopidogrel (PlavixÒ), other antiplatelet agents) or anticoagulants (heparin, low molecular weight heparin, warfarin, lepirudin, or other anticoagulants) and inability to temporarily hold such medications for endoscopy.
* Decompensated disease (e.g., active angina, unstable angina, or MI within two months, congestive heart failure, renal failure and dialysis, respiratory insufficiency with FEV1 < 1L or oxygen dependence, cirrhosis, uncontrolled diabetes)
* Ongoing substance abuse
* Receipt of a non-HIV vaccine within 30 days
* Opportunistic infection within 60 days
* Immunosuppressive medications (e.g., systemic corticosteroids, tacrolimus, sirolimus, mycophenolate, azathioprine, interferon, and cancer chemotherapy) within 60 days
* Alcoholism including binging
* history of clinically significant medical disease, includes renal (creatinine >2 mg/dL), liver (documented cirrhosis based on histology or ALT/AST greater than 2 1/2 times normal), cardiac failure (NY classification III/IV), or uncontrolled diabetes (Hgb- A1c>8%).
* Regular use of NSAIDs (daily more than three days a week during the prior two weeks of starting the study)
* Antibiotic use during prior four weeks to the colonoscopy).
* Abnormal blood clotting time (e.g., prolonged PT) or use of anticoagulant during 3-7 days prior to colonoscopy that would preclude biopsy sample collection.
* Obesity (BMI>30 because it can affect the microbiota community.
* Use of special diet like vegan, vegetarian, gluten-free, Paleo, specific carbohydrate diet because these diets can impact the microbiota community.
* Inflammatory bowel disease.
* Celiac disease.
* GI cancers
* gastrointestinal surgeries/resection
* Inability to sign an informed consent form.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Sugar test for intestinal permeability after prebiotic consumption in substudy | 10 days
  Measure the permeation of sugar probes following an oral test dose of sugars as this is standard for evaluating intestinal barrier integrity

SECONDARY OUTCOMES:
Change in stool and intestinal microbiota composition after prebiotic consumption | 10 days
  A combination of 16S rRNA gene amplicon sequencing and shotgun metagenome sequencing will be used to characterize microbial community structure in intestinal biopsies and stool.
Change in plasma and stool SCFA level before and after prebiotic treatment | 10 days
  Mass spectrometry and NMR

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Keshavarzian, Chicago, IL 60612, Illinois, United States